CLINICAL TRIAL: NCT04759638
Title: Body Mass Index Role in the Oncological Outcome of Locally Advanced Rectal Cancer: The Two BMI Extremes as Comparative Groups, A Retrospective Study
Brief Title: Short Running Head Obesity in Rectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: King Hussein Cancer Center (Other)
Responsible Party: Principal Investigator, Mahmoud Al-Masri, Chairman, Department of Surgery, King Hussein Cancer Center
Other Study IDs: 17KHCC42
Record Dates: First submitted 2021-02-08; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Rectal Cancer
Keywords: Oncology; Colorectal Cancer; Surgery; Surgical Oncology; Obesity
MeSH Terms: conditions — Rectal Neoplasms; Neoplasms; Colorectal Neoplasms; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rectal Cancer: Rectal Cancer

SUMMARY:
There is a controversy regarding the effect of the two Body Mass Index (BMI) extremes on the oncological outcome of rectal cancer.

The obesity paradox appears to exist in rectal cancer patients treated with nCRT and surgery, as it was associated with significantly higher rates of pathological complete response and R0 resection.

Underweight patients were at higher risk for anastomotic leak and R1 resection.

DETAILED DESCRIPTION:
Background:

Obesity and underweight are associated with increased risk of postoperative morbidity in colorectal cancer patients undergoing surgery. There is a controversy regarding the effect of the two Body Mass Index (BMI) extremes on the oncological outcome of rectal cancer.

Objective:

The aim of this study was to evaluate the effect of BMI on short- and long-term oncological outcomes as well as postoperative complications in rectal cancer patients who received neoadjuvant chemoradiotherapy (nCRT) followed by surgery.

Setting:

Tertiary Cancer Center serving pediatric and adult patients in Jordan and the Middle East.

Patients:

The medical records of patients with stage II-III rectal cancer who received nCRT followed by surgery during 2006 to 2018 were retrospectively reviewed. The patients were subdivided according to their BMI into less than 20 kg/m2 defined as underweight; between 20 to 30 kg/m2 defined as normal range weight, above 30 kg/m2 defined as obese.

Main Outcome Measures:

Disease-Free Survival (DFS), Overall Survival, Pathological Complete Response (CR)

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent rectal surgery at King Hussein Cancer Center (KHCC) from 2006 to 2018 were identified. Those with locally advanced rectal cancer (stages II and III) who underwent nCRT followed by surgery with curative intent were included.

Exclusion Criteria:

* Patients with early rectal cancer (stage I) who did not require nCRT and those who underwent rectal surgery as part of a staged or simultaneous approach for metastatic disease (stage IV) were excluded.

Age Groups: Child, Adult, Older Adult
Study Population: 294 patients included in the study
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | 5 yers
  Disease-free survival (DFS) was defined as the time from surgical resection to disease recurrence (including loco-regional failure or metastases) or death of any cause
Overall Survival (OS) | 5 years
  Overall survival (OS) was defined as the time interval from surgical resection to either death from any cause or last follow up

SECONDARY OUTCOMES:
Pathological Complete Response (CR) | 5 years
  Pathological CR was defined as no viable cancer cells in the excised specimen.

CONTACTS AND LOCATIONS:
Locations (1):
- King Hussein Cancer Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No